CLINICAL TRIAL: NCT00727558
Title: A Comparison of Daily Disposable Contact Lenses.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: Visioncare Research Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0808; PROD-501
Record Dates: First submitted 2008-07-30; First posted 2008-08-04 (Estimated); Results first posted 2010-02-18 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Myopia
Keywords: refractive error
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- narafilcon A (Active Comparator): spherical soft contact lens worn as a daily disposable modality for one week
  Interventions: Device: narafilcon A
- nelfilcon A (Active Comparator): spherical soft contact lens worn as a daily disposable modality for one week
  Interventions: Device: nelfilcon A; Device: narafilcon A

INTERVENTIONS:
Device: nelfilcon A — spherical soft contact lens
  Arms: nelfilcon A
Device: narafilcon A — spherical soft contact lens

SUMMARY:
This study seeks to evaluate the clinical performance of a new CE marked daily disposable contact lens that contains a wetting agent to a recently improved daily disposable contact lens.

ELIGIBILITY:
Inclusion Criteria:

* They are of legal age (18 years) and capacity to volunteer.
* They understand their rights as a research subject and are willing to sign a Statement of Informed Consent.
* They are willing and able to follow the protocol.
* They would be expected to attain at least 6/9 (20/30) in each eye with the study lenses.
* They are able to wear contact lenses with a back vertex power of -1.00 to -6.00DS.
* They have a maximum of 1.00D of refractive astigmatism (i.e. ≤ 1.00 DC).
* They have successfully worn contact lenses within six months of starting the study.

Exclusion Criteria:

* They have an ocular disorder which would normally contra-indicate contact lens wear.
* They have a systemic disorder which would normally contra-indicate contact lens wear.
* They are using any topical medication such as eye drops or ointment.
* They are aphakic.
* They have had corneal refractive surgery.
* They have any corneal distortion resulting from previous hard or rigid lens wear or has keratoconus.
* They are pregnant or lactating.
* They have grade 2 or greater of any of the following ocular surface signs: corneal oedema, corneal vascularisation, corneal staining, tarsal conjunctival changes or any other abnormality which would normally contraindicate contact lens wear.
* They have any infectious disease (e.g. hepatitis) or any immunosuppressive disease (e.g. HIV).
* They have diabetes.
* They have taken part in any other clinical trial or research, within two weeks prior to starting this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 248 (Actual)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United Kingdom (19):
  - Ellis & Killpartrick, Bath, Bath
  - Simon Donne Opticians 3-4, Bedford, Bedfordshire
  - Brock & Houlford, Brislington, Bristol
  - The Contact Lens Centre, Plymouth, Devon
  - Keith Tempany Opticians, Broadstone, Dorset
  - Eyecare, Ilford, Essex
  - Leightons Opticians, Albans, Herts
  - Hazel Smith Opticians, Shanklin, Isle of Wight
  - Bowden & Lowe, Gillingham, Kent
  - David Gould Opticians, Rawtenstall, Lancashire
  - Vision Express Optical Lab, Hendon, London
  - Hawkes & Wainer, London, London
  - City Opticians, London, London
  - David H Burns BSC, FCOptom, Tottenham, London
  - First Contact Opticians, Eastcote Pinner, Middlesex
  - Tompkins Knight & Son, Northampton, Northampton
  - Chalmers & Son (Opticians), Cardiff, South Glamorgan
  - Susan R Bowers Opticians, Coventry, West Midlands
  - Viewpoint, York, York

RESULTS

PARTICIPANT FLOW:
Groups:
- Narafilcon A; Nelfilcon A: soft contact lens worn as a daily disposable modality for one week
Period: Overall Study
Arm/Group | Narafilcon A | Nelfilcon A
Started | 127 | 121
Completed | 125 | 118
Not Completed | 2 | 3
Not completed — Lens issue | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Subject unable to return for follow-up | 1 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Narafilcon A | Nelfilcon A | Total
Number analyzed (Participants) | 125 | 118 | 243
Age, Continuous [Mean (Standard Deviation); unit: years] — Includes completed subjects only
  years | 33.0 (9.5) | 32.9 (10.6) | 33.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Includes completed subjects only
  Participants
    Female | 90 | 92 | 182
    Male | 35 | 26 | 61
Region of Enrollment [Number; unit: participants] — Includes completed subjects only
  participants
    United Kingdom | 125 | 118 | 243

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort
Description: Single question: Comfort scale: 0=N/A, 1=Poor, 2=Fair, 3=Good, 4=Very Good, 5=Excellent
Time Frame: at 1 week of wear.
Population: Analysis includes participants who completed the protocol and had no missing data (n=240)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Narafilcon A | Nelfilcon A
Number analyzed (Participants) | 124 | 116
Units on a scale | 3.903 (0.1446) | 3.349 (0.1389)
Statistical Analysis 1: Comparison: Narafilcon A vs Nelfilcon A; Alternative hypothesis: narafilcon A is superior to nelfilcon A; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.554, 97.47% CI [0.1721 to 0.554], Standard Error of Mean 0.1943 — The mean difference is narafilcon A minus nelfilcon A

2. Primary Outcome: Measured Limbal Hyperemia
Description: Measurement of redness of the limbus, graded using half-grade increments using the following scale: 0=none, 1=trace, 2=mild, 3=moderate, 4=severe.
Time Frame: at 1 week of wear.
Population: Analysis includes participants who completed the study per protocol and had no missing data (n=243).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Narafilcon A | Nelfilcon A
Number analyzed (Participants) | 125 | 118
Units on a scale | 0.364 (0.05494) | 0.5374 (0.0558)
Statistical Analysis 1: Comparison: Narafilcon A vs Nelfilcon A; Alternative hypothesis: narafilcon A is superior to nelfilcon A; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.1734, 97.47% CI [-0.1734 to -0.1037], Standard Error of Mean 0.03555 — Mean difference is narafilcon A minus nelfilcon A

3. Secondary Outcome: Overall Handling
Description: Rating of overall ease of handling using the following scale: 0=N/A, 1=Poor, 2=Fair, 3=Good, 4=Very Good, 5=Excellent.
Time Frame: at 1 week of wear
Population: Analysis includes participants who completed the study per protocol and had no missing data (n=240).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Narafilcon A | Nelfilcon A
Number analyzed (Participants) | 124 | 116
Units on a scale | 4.0959 (0.1209) | 3.6991 (0.1172)
Statistical Analysis 1: Comparison: Narafilcon A vs Nelfilcon A; Alternative hypothesis: narafilcon A is superior to nelfilcon A; Test type: Superiority or Other; Mixed Models Analysis; Median Difference (Final Values) = 0.3968, 98.7% CI [0.04983 to 0.3968], Standard Error of Mean 0.1548 — The mean difference is narafilcon A minus nelfilcon A

4. Secondary Outcome: How Comfortable Eyes Feel at the End of the Day
Description: Rating of "How comfortable did your eyes feel at the end of the day when wearing the contact lenses provided" using the following scale: 1=extremely uncomfortable, 2= very uncomfortable, 3=slightly uncomfortable, 4=comfortable, 5=very comfortable.
Time Frame: at 1 week wear
Population: Analysis includes participants who completed the study per protocol and had no missing data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Narafilcon A | Nelfilcon A
Number analyzed (Participants) | 124 | 116
Units on a scale | 3.8669 (0.1546) | 3.4794 (0.1487)
Statistical Analysis 1: Comparison: Narafilcon A vs Nelfilcon A; Alternative hypothesis: narafilcon A is superior to nelfilcon A; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.3875, 98.7% CI [0.03714 to 0.3875], Standard Error of Mean 0.2054 — The mean difference is narafilcon A minus nelfilcon A

5. Secondary Outcome: End of Day Comfort
Description: Rating of comfort at the end of the day using the following scale: 0=N/A, 1=Poor, 2=Fair, 3=Good, 4=Very Good, 5=Excellent
Time Frame: at 1 week of wear
Population: Analysis includes participants who completed the study per protocol and had no missing data (n=240).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Narafilcon A | Nelfilcon A
Number analyzed (Participants) | 124 | 116
Units on a scale | 3.425 (0.129) | 2.7515 (0.1269)
Statistical Analysis 1: Comparison: Narafilcon A vs Nelfilcon A; Alternative hypothesis: narafilcon A is superior to nelfilcon A; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.6735, 98.7% CI [0.213 to 0.6735], Standard Error of Mean 0.1563 — The mean difference is narafilcon A minus nelfilcon A

6. Secondary Outcome: Initial Comfort
Description: Rating of "comfort immediately when you first put them on" using the following scale: 0=N/A, 1= Poor, 2=Fair, 3=Good, 4=Very Good, 5=Excellent.
Time Frame: at 1 week
Population: Analysis includes participants who completed the study per protocol and had no missing data (n=240).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Narafilcon A | Nelfilcon A
Number analyzed (Participants) | 124 | 116
Units on a scale | 4.0306 (0.1352) | 3.8986 (0.1312)
Statistical Analysis 1: Comparison: Narafilcon A vs Nelfilcon A; Alternative hypothesis: narafilcon A is superior to nelfilcon A; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.132, 98.7% CI [-0.2375 to 0.132], Standard Error of Mean 0.1648 — Mean difference is narafilcon A minus nelfilcon A

7. Secondary Outcome: Inferior Region Corneal Staining
Description: National Eye Institute (NEI) 0-3 scale: grade 0=normal, grade 1=mild, grade 2=moderate, grade 3=severe.
Time Frame: at 1 week of wear
Population: Analysis includes participants who completed the study per protocol and had no missing data (n=243).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Narafilcon A | Nelfilcon A
Number analyzed (Participants) | 125 | 118
Units on a scale | 0.311 (0.03884) | 0.5579 (0.03974)
Statistical Analysis 1: Comparison: Narafilcon A vs Nelfilcon A; Alternative hypothesis: narafilcon A is superior to nelfilcon A by having a lower level of inferior region corneal staining; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.2469, 97.47% CI [-0.2469 to -0.1599], Standard Error of Mean 0.04448 — The mean difference is narafilcon A minus nelfilcon A

ADVERSE EVENTS:
Arm/Group | Narafilcon A | Nelfilcon A
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/121
Other Adverse Events (participants affected / at risk) | 0/127 | 0/121

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish, divulge, reveal, disclose, or use the data and or results of the study without prior written consent of Vistakon.